CLINICAL TRIAL: NCT00440336
Title: Comparison of Efficacy of Prostaglandin Analogues (Xalatan) and Aqueous Suppressants (Cosopt) in Reducing Intraocular Pressure Following Selective Laser Trabeculoplasty in the Management of Open-Angle Glaucoma.
Brief Title: Comparison of Efficacy of Two Groups of Glaucoma Drops (Xalatan vs.Cosopt) in Reducing Eye Pressure Following Laser (SLT)Treatment in the Management of Glaucoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advanced Glaucoma Specialists (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 31663
Record Dates: First submitted 2007-02-24; First posted 2007-02-27 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Open Angle Glaucoma
Keywords: IOP; SLT; Laser; Cosopt
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — dorzolamide-timolol combination; Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cosopt
Drug: Xalatan

SUMMARY:
WHAT IS THIS STUDY ABOUT? Glaucoma and ocular hypertension are chronic eye diseases that can damage the optic nerve and lead to vision loss or blindness. The optic nerve acts like an electric cable with over a million wires. This nerve is responsible for carrying images from the eye to the brain. The way glaucoma and ocular hypertension cause blindness depends on many factors, but the most important factor is the increased pressure inside the eye (intraocular pressure).

There is no cure for glaucoma or ocular hypertension. However, lowering the pressure inside the eye has been shown to slow the progression of disease. Intraocular pressure can be lowered by glaucoma medication, laser treatment, or surgery.

You have open angle glaucoma, pseudoexfoliative glaucoma, or ocular hypertension. Researchers want to find out more about how 2 drugs called Cosopt (dorzolamide hydrochloride and timolol maleate) and Xalatan (latanoprost) can help people with these conditions.

Cosopt and Xalatan are both eye drops that are approved by the U.S. Food and Drug Administration (FDA) to reduce intraocular pressure in people with open angle glaucoma and ocular hypertension.

The study doctor will do a laser procedure called Selective Laser Trabeculoplasty (SLT) on people in this study to help lower their intraocular pressure. The FDA has approved SLT to treat open angle glaucoma and ocular hypertension.

Then the study doctor will ask some participants to use either Cosopt or Xalatan, if their intraocular pressure is still too high 4 to 6 weeks after the SLT procedure. The study doctor wants to see which of the 2 study drugs (Cosopt or Xalatan) is better at reducing intraocular pressure after SLT.

It is planned that about 30 people with glaucoma or ocular hypertension who are at least 18 years old will be in this study. Out of the participants whose intraocular pressure is still too high after SLT, half will use Cosopt and half will use Xalatan. You do not have to be in this study to have SLT or to use Cosopt or Xalatan.

DETAILED DESCRIPTION:
Introduction Selective Laser Trabeculoplasty has been shown as a relatively safe and effective treatment modality for lowering IOP in various forms of open-angle glaucoma (Latina et al). It lowers IOP by increasing aqueous outflow through its effect at cellular level possibly either (1) through migration and phagocytosis of trabecular meshwork debris by macrophages or (2) by stimulating the proliferation of healthy trabecular and endothelial cells.

Cases who don't achieve target IOP following SLT therapy need additional treatment in form of topical medications. Conventionally common topical antiglaucoma medications to treat glaucoma after SLT therapy either suppress aqueous secretion (B-blockers or carbonic anhydrase inhibitors) or enhances uveoscleral aqueous outflow (Prostaglandin analogues). Since Selective Laser Trabeculoplasty acts on outflow pathway, further additional IOP reduction can be achieved more effectively by a class of drug which acts on different pathway; on aqueous secretion by aqueous suppressants like Cosopt. In contrast drugs acting on outflow pathway like prostaglandin analogue ( Xalatan etc) will possibly be less additive in further reducing IOP after SLT since SLT also has effect on the same pathway- outflow pathway.

Previous studies (Fechtner et al. J Ocul Pharmacol Ther. 2005 Jun;21(3):242-9 and Fechtner et al. Acta Ophthalmol Scand. 2004 Feb;82(1):42-8.) have shown equal efficacy of Cosopt and Latanoprost in reducing IOP in treatment of glaucoma. But to our knowledge, no long term prospective study has evaluated aqueous suppressants (Cosopt) and prostaglandin analogues with respect to their comparative efficacy in treatment of uncontrolled glaucoma status post SLT therapy.

OBJECTIVE The primary objective of this study is to compare the IOP lowering efficacy of aqueous suppressants (Cosopt) and prostaglandin analogues (Xalatan) when used status post SLT in the management of Open Angle Glaucoma or Ocular Hypertension.

INCLUSION CRITERIA 1. Adult subjects of either sex, of any race, eighteen years of age or older. 2 Diagnosis: Primary Open Angle Glaucoma, Pseudoexfoliation Glaucoma, Ocular Hypertension.

3. Mild to moderate glaucoma only: Pattern standard deviation (PSD); more than 1DB and less than 6 DB on Humphrey Visual Field.

3. Subject may be;

* A newly diagnosed glaucoma or
* A pre-existing glaucoma on not more than two topical antiglaucoma medications. 3 On no systemic medications known to increase IOP (e.g. steroids) 4 Visual acuity equal or better than 20/200 in the study eye 5. IOP less than 35 mm Hg in the study eye 6 No previous intraocular surgery within last 6 months, except laser PI greater than 3 months ago.

EXCLUSION CRITERIA Pigmentary OAG, Proliferative diabetic retinopathy, History of chronic or recurrent severe inflammatory eye disease (i.e. scleritis, uveitis, herpes keratitis), known allergy to COSOPT or any of Prostaglandin Analogues, Chronic Obstructive Airways Disease (COPD), sinus bradycardia (heart rate < 60 beats per minute), second or third-degree atrioventricular block, overt cardiac failure. Pregnant and nursing mothers.

STUDY DESIGN: Single site, unmasked, prospective, randomized study STUDY PROCEDURE

Visit 1 Visit 2 Visit 3 Visit 4 Visit 5 Visit 6 Screening Phase SLT Treatment Phase Safety check 2 weeks after SLT RANDOMIZATION 4 to 6 weeks after SLT Follow up visit, 6 weeks after randomization Last Visit 3 months after randomization Determine eligibility by doing routine eye exam including IOP check by Goldmann applanation tonometer, Gonioscopy, fundus exam, Humphrey Visual Field (if HVF not done within last 6 months).

Subjects, who fulfill the eligibility criteria and give consent for participating in study, will be scheduled for SLT. All eligible subjects will receive SLT. Pre-existing glaucoma cases already on antiglaucoma medications will discontinue all the antiglaucoma medications since the day of SLT treatment and will be off the drops for next 4 to 6 weeks. Similarly newly diagnosed glaucoma will not be on any antiglaucoma medications. for next 4 to 6 weeks. Each subject will have IOP check at 2 weeks after SLT treatment. It will be done to rule out any unusual IOP spike following SLT. Each subject will have routine eye exam including IOP check at this visit. The subjects with uncontrolled IOP despite SLT therapy will be randomized to receive either COSOPT or Prostaglandin analogue (XALATAN). IOP check and routine eye exam. IOP check, routine eye exam including fundus exam and Humphrey Visual Field.

 If IOP is uncontrolled at the visit 5, a stepped drug therapy will be initiated based on following protocol:

1. For patients who are in Cosopt group after randomization. Sequence of additional medications will be following:

   First Step: Alphagan (Brimonidine) Second Step: Prostaglandin Analogues
2. For patients who are in Xalatan group after randomization. Sequence of additional medications will be following:

First Step: Alphagan (Brimonidine) Second Step: Dorzolamide (Trusopt)

Note: IOP will be measured using a Goldmann Applanation Tonometer at 8 AM and 10 AM at visits: Visit I, Visit IV, Visit V and Visit VI. A ± 30 minute window will be allowed for each measurement recording.

IOP measurement at Visit II (SLT treatment phase) and Visit III (safety check) can be done at random time.

Duration of Study Participation; Subjects who are eligible to participate in the study shall be enrolled for approximately 6 months. References; Fechtner RD, McCarroll KA, Lines CR, Adamsons IA. Efficacy of the dorzolamide/timolol fixed combination versus latanoprost in the treatment of ocular hypertension or glaucoma: combined analysis of pooled data from two large randomized observer and patient-masked studies.J Ocul Pharmacol Ther. 2005 Jun;21(3):242-9 Fechtner RD, Airaksinen PJ, Getson AJ, Lines CR, Adamsons IA; COSOPT versus XALATAN Study Groups.

Efficacy and tolerability of the dorzolamide 2%/timolol 0.5% combination (COSOPT) versus 0.005% (XALATAN) in the treatment of ocular hypertension or glaucoma: results from two randomized clinical trials. Acta Ophthalmol Scand. 2004 Feb;82(1):42-8.

Latina MA, Tumbocon Ja. SLT: a new treatment option for open-angle glaucoma. Curr Opin Ophthalmol 2002; 13:94-6

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects of either sex, of any race, eighteen years of age or older.
2. Diagnosis: Primary Open Angle Glaucoma, Pseudoexfoliation Glaucoma, Ocular Hypertension.
3. Mild to moderate glaucoma only: Pattern standard deviation (PSD); more than 1DB and less than 6 DB on Humphrey Visual Field.
4. Subject may be:

   * A newly diagnosed glaucoma or
   * A pre-existing glaucoma on not more than two topical antiglaucoma medications.
5. On no systemic medications known to increase IOP (e.g. steroids)
6. Visual acuity equal or better than 20/200 in the study eye
7. IOP less than 35 mm Hg in the study eye
8. No previous intraocular surgery within last 6 months, except laser PI greater than 3 months ago.

Exclusion Criteria:

1. Pigmentary OAG,
2. Proliferative diabetic retinopathy,
3. History of chronic or recurrent severe inflammatory eye disease (i.e. scleritis, uveitis, herpes keratitis),
4. Known allergy to COSOPT or any of Prostaglandin Analogues,
5. Chronic Obstructive Airways Disease (COPD),
6. Sinus bradycardia (heart rate < 60 beats per minute),
7. Second or third-degree atrioventricular block,
8. Overt cardiac failure.
9. Pregnant and nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-10

PRIMARY OUTCOMES:
Reduction in Intraocular Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mark Latina, Principal Investigator — Advanced Glaucoma Specialist
Locations (1):
- Advanced Glaucoma Specialist, Reading, Massachusetts, United States